CLINICAL TRIAL: NCT00100594
Title: A Feasibility Study of Lamivudine/Zidovudine (3TC/ZDV) Plus Efavirenz (EFV) as Initial Therapy of HIV-1 Infected Patients in a Rural Area of China
Brief Title: Efavirenz and Lamivudine/Zidovudine for Treatment-Naive HIV Infected People in Wenxi County, Shanxi Province, China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIPRA CH 004
Record Dates: First submitted 2005-01-03; First posted 2005-01-04 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: HIV Infections
Keywords: Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — efavirenz; lamivudine, zidovudine drug combination

INTERVENTIONS:
Drug: Efavirenz
Drug: Lamivudine/zidovudine

SUMMARY:
The purpose of this study is to determine the safety, effectiveness, and tolerability of the anti-HIV drugs efavirenz and lamivudine/zidovudine given to treatment-naive HIV infected people in Wenxi County, Shanxi Province, China.

DETAILED DESCRIPTION:
HIV infection in China has reached epidemic proportions, especially in poor rural communities. Among the infected are former commercial plasma donors who became infected through contaminated blood collection equipment. This study will evaluate the safety, efficacy, and tolerability of an antiretroviral (ARV) regimen given to treatment-naive HIV infected adults. Participants will be recruited in Wenxi County, Shanxi Province.

This study will last 1 year. At study entry, all study participants will be given an ARV regimen consisting of lamivudine/zidovudine twice daily and efavirenz once daily. There will be 11 study visits; a physical exam, blood collection, and vital signs measurement will occur at all study visits. Participants will also receive safe sex and adherence counseling at all visits. Participants will be asked to complete an adherence questionnaire and will have their pills counted at most visits.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* Antiretroviral naive
* CD4 count of less than 350 cells/mm3 within 30 days of study entry
* Willing to use acceptable forms of contraception
* Willing to stay in the study area for the duration of the study
* Willing to not consume traditional Chinese medicines for the duration of the study
* Willing to adhere to the follow-up study schedule

Exclusion Criteria:

* Presence of an acute serious medical illness within 14 days prior to study entry. Participants with recently diagnosed opportunistic infections (except tuberculosis [TB]) and are stable on therapy for more than 30 days are eligible.
* Current pancreatitis
* Require certain medications
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-05; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Cumulative treatment failure at 52 weeks, defined by virologic failure or all-cause mortality
treatment-limiting toxicity, defined by any participant in whom treatment is permanently discontinued according to toxicity guidelines

SECONDARY OUTCOMES:
Tolerability, defined by premature discontinuation or failure to take ARV regimen for more than 8 consecutive weeks
adherence, defined by continuous and dichotomous measure
ARV drug resistance

CONTACTS AND LOCATIONS:
Overall Officials: Yunzhen Cao, MD, Study Chair — The AIDS Research Center, Chinese Academy of Medical Sciences, Peking Union Medical College

REFERENCES:
- [Background] Wu Z, Rou K, Cui H. The HIV/AIDS epidemic in China: history, current strategies and future challenges. AIDS Educ Prev. 2004 Jun;16(3 Suppl A):7-17. doi: 10.1521/aeap.16.3.5.7.35521. PMID 15262561